CLINICAL TRIAL: NCT00778245
Title: An Open - Label, Comparative, Randomized, Single-Dose, 2-Way Crossover Bioavailability Study of Ranbaxy and Bristol-Myers Squibb Company (CEFZIL ®) 500 mg Cefprozil Tablets in Healthy Adult Volunteers Under Fed Conditions.
Brief Title: Bioequivalence Study of Cefprozil Tablets, USP 500 mg Undef Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AA27169
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence cefprozil 500mg tablets fed conditions
MeSH Terms: interventions — Cefprozil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): cefprozil 500mg tablets of Ranbaxy
  Interventions: Drug: cefprozil 500mg tablets
- 2 (Active Comparator): CEFZIL ® 500 mg tablets of Bristol-Myers Squibb Company, USA
  Interventions: Drug: cefprozil 500mg tablets

INTERVENTIONS:
Drug: cefprozil 500mg tablets

SUMMARY:
The objective of this study is to assess the single - dose relative bioavailability of Ranbaxy and Bristol-Myers Squibb Company (CEFZIL ®) 500 mg cefprozil tablets, under fed conditions.

DETAILED DESCRIPTION:
A single dose, randomized, two-period, two-treatment, two-sequence crossover study design was used to evaluate the relative bioavailability of the cefprozil tablet products when dosed (1 x 500 mg) under fed conditions. The washout period will be at least 14 days between doses.

Twenty four plus two alternate (24 + 2) subjects were enrolled in this study and all volunteers were healthy adults. Twenty six (24 + 2) subjects began the study, and twenty-five (23 + 2) subjects completed the clinical portion of the study in its entirety.

ELIGIBILITY:
Inclusion Criteria:

* Subject candidates must fulfill all of the following inclusion criteria t be eligible for participation in the study, unless otherwise specified:

  1. Healthy adult male or female volunteers, 18 to 55 years of age
  2. Weighing at least 52 kg for males and 45 kg for females and within 15% of their ideal weights (table of 'Desirable Weights of Adults', Metropolitan Life Insurance Company, 1983)
  3. Medically healthy subjects with clinically normal laboratory profiles and ECGs
  4. Females of child bearing potential should either be sexually inactive (abstinent) for 14 days prior to the first dose and throughout the study or be using one of the following acceptable birth control methods:
* Surgically sterile (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) 6 months minimum
* IUD in place for at least 3 months
* Barrier methods (condom, diaphragm) with spermicide for at least 14 days prior to the first dose and throughout the study
* Surgical sterilization of the partner (vasectomy for 6 months minimum)
* Hormonal contraceptives for at least 3 months prior to the first dose of the study
* Other birth control methods may be deemed acceptable e) Post menopausal women with amenorrhea for at least 2 years will be eligible f) Voluntarily consent to participate in the study

Exclusion Criteria:

* Subject candidates must not be enrolled in the study if they meet any of the following criteria:

  1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
  2. In addition, history or presence of:
* alcohol or drug abuse within the past year
* hypersensitivity or idiosyncratic reaction to cefprozil, other cephalosporin antibiotics, or penicillin c) Female subjects who are pregnant or lactating d) Subjects who have been on a special diet (for whatever reason) during the 28 days prior to the first dose and throughout the study e) Subjects who through completion of the study, would have donated in excess of:
* 500 mL of blood in 14 days
* 1500 mL of blood in 180 days
* 2500 mL of blood in 1 year f) Subjects who have participated in another clinical trial within 28 days prior to the first dose.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2005-05; Primary Completion 2005-06 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- MDS Pharma Services, Montreal, Quebec, Canada

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html